CLINICAL TRIAL: NCT04765956
Title: Intravascular Identification and Drug-Eluting Balloon Treatment of Vulnerable Lipid-Rich Plaques
Acronym: DEBuT-LRP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, J.P.S Henriques, Prof. Dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEBuT-LRP
Record Dates: First submitted 2021-02-18; First posted 2021-02-23 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Coronary Artery Disease
Keywords: Lipid-rich plaque; Non-ST-elevation myocardial infarction; Near-infrared spectroscopy; Drug-eluting balloon
MeSH Terms: conditions — Coronary Artery Disease; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: Prospective single-arm clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Drug-eluting balloon treatment (Experimental): Drug-eluting balloon (DEB) treatment of lipid-rich plaque
  Interventions: Device: Drug-eluting balloon treatment

INTERVENTIONS:
Device: Drug-eluting balloon treatment — Drug-eluting balloon (DEB) treatment of lipid-rich plaque

SUMMARY:
Rationale: Two-thirds of intracoronary thrombi causing acute coronary syndrome (ACS) result from rupture of lipid-rich plaques (LRP). After treatment of the culprit lesion in ACS patients, additional LRPs are found in approximately 50% of patients. Near infrared spectroscopy (NIRS) combined with intracoronary ultrasound (IVUS) can identify these vulnerable plaques during coronary angiography (CAG) and is able to assess plaque characteristics and the lipid-core burden index in a 4mm segment (LCBImm4). It is currently unknown whether treatment of LRPs leads to plaque stabilization, potentially reducing the number of subsequent ACS. We hypothesize that LRPs can be treated with balloons coated with an antiproliferative drug (i.e. drug-eluting balloons; DEB) to deliver selective pharmacotherapeutic treatment to halt the local atherosclerotic process and subsequently reduce the risk for atherosclerotic events.

Objectives: To determine the change in plaque characteristics of non-culprit LRPs, as measured with IVUS/NIRS, after treatment with DEB in patients with ACS.

Study design: Prospective single-arm clinical trial

Study population: Patients with non-ST-elevation acute coronary syndromes

Intervention: If a LRP is detected with IVUS/NIRS, it will be treated with DEB. In case multiple LRPs are detected, only one will be treated.

Main study endpoints: The difference in LCBImm4 between baseline and 9 months of plaques treated with DEB.

ELIGIBILITY:
Inclusion Criteria:

* Patient has an acute coronary syndrome without ST-segment elevation on the ECG (NSTE-ACS), including non-ST-elevation myocardial infarction and unstable angina pectoris, defined according to the Fourth Universal Definition of Myocardial Infarction.
* An invasive revascularization strategy for NSTE-ACS with PCI is chosen.

Exclusion Criteria:

- Angiographic exclusion criteria:

1. Previous coronary artery bypass-grafting;
2. Presence of a chronic total occlusion;
3. Too many (complex) coronary lesions requiring staged PCI procedure(s);
4. Procedural complication of the index PCI;

   - Clinical exclusion criteria:
5. Unstable patients (the presence of cardiogenic shock, need for intubation, need for inotropes);
6. Patients with ST-segment elevations on the ECG requiring immediate primary PCI;
7. Body weight > 250 kg;
8. Known renal insufficiency (estimated Glomerular Filtration Rate [eGFR] <30 mL/min/1.73m2 or subject on dialysis);
9. Hypersensitivity or allergy to contrast with inability to properly pre-hydrate;
10. Presence of a comorbid condition with a life expectancy of less than one year;
11. Participation in another trial;
12. Subject is belonging to a vulnerable population (per investigator's judgment, e.g., subordinate hospital staff) or is unable to read or write.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-19 (Actual); Primary Completion 2023-09-09 (Estimated); Study Completion 2023-09-09 (Estimated)

PRIMARY OUTCOMES:
LCBImm4 difference of DEB-treated LRPs | 9 months
  The difference in LCBImm4 between baseline and 9 months follow-up of lipid-rich plaques treated with drug-eluting balloon, as measured with near-infrared spectroscopy (NIRS).

SECONDARY OUTCOMES:
The change in lipid-core burden index in a 4 mm segment (LCBImm4) as measured with IVUS + NIRS from baseline to 9 month follow-up in identified additional LRPs that are not treated with DEB. | 9 months
Rate of flow-limiting dissections necessitating bail-out stent implantation; | 9 months
Rate of periprocedural myocardial infarction; | 9 months
Rate of LRP lesion failure (defined as cardiac death, myocardial infarction, or ischemia-driven revascularization related to an identified non-culprit LRP lesion up to one-year follow-up); | 1 year
Patient-oriented composite outcomes, defined as all-cause mortality, myocardial infarction, or any repeat revascularization up to one-year follow-up; | 1 year
Additional IVUS + NIRS lesion characteristics: plaque volume | 9 months
Additional IVUS + NIRS lesion characteristics: minimal lumen area | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, location AMC, Amsterdam, Netherlands